CLINICAL TRIAL: NCT04666259
Title: An Open Label, Multi-center Phase IIIb Study of Asciminib (ABL001) Monotherapy in Previously Treated Patients With Chronic Myeloid Leukemia in Chronic Phase (CML-CP) With and Without T315I Mutation
Brief Title: Asciminib in Monotherapy for Chronic Myeloid Leukemia in Chronic Phase (CML-CP) With and Without T315I Mutation
Acronym: AIM4CML
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CABL001AUS04
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Results first posted 2024-07-12 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Chronic Myelogenous Leukemia - Chronic Phase
Keywords: CML; T315I mutation; CP; Asciminib,; BCR-ABL,; ABL001,; CML-AP,; ELN; MMR; Molecular Response; MR4.5; MR4; RQ-PCR; AIM4CML,; tyrosine Kinase Inhibitor; TKI; adult
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — asciminib

STUDY DESIGN:
Masking Description: Cohort A and B will be randomized but not C
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): 40 mg asciminib orally twice daily (BID)
  Interventions: Drug: ABL001
- Cohort B (Experimental): 80 mg asciminib orally once daily (QD)
  Interventions: Drug: ABL001
- Cohort C (Experimental): 200 mg asciminib orally twice daily (BID)
  Interventions: Drug: ABL001

INTERVENTIONS:
Drug: ABL001 — Asciminib will be supplied as 20 mg or 40 mg strength tablets will be administered orally in accordance with the assigned cohort.

SUMMARY:
This study was a multicenter Phase IIIb open-label, three-cohort study of asciminib in patients with CML-CP without T315I mutation who have had at least 2 prior TKIs and CML-CP harboring the T315I mutation with at least 1 prior TKI

DETAILED DESCRIPTION:
This trial consisted of three periods: screening and baseline for up to 21 days, active treatment for up to 72 weeks and a safety follow up period for 30 days.

One hundred and fifteen (115) patients with chronic myeloid leukemia in chronic phase (CML-CP) without T315I mutation who have had at least 2 prior Tyrosine Kinase Inhibitors (TKIs) and CML-CP with the T315I mutation with at least 1 prior TKI were planned for this study, however the study was finally completed with 56 participants due to enrollment issues.

Informed consent was obtained before any procedures were performed for the study including eligibility assessments. The results of the real time quantitative polymerase chain reaction (RQ-PCR) must be available prior to randomization and first dose of study treatment.

Patients with CML-CP without T315I mutation were randomly assigned to either cohort A or B. Patients with the T315I mutation were enrolled in cohort C. During treatment period asciminib was taken orally: Cohort A was administered 40 mg twice a day, Cohort B was administered 80 mg once a day and Cohort C was administered 200 mg twice a day. The patients were treated up to end of study treatment period defined as up to 72 weeks after the last patient receives the first dose. Patients may have been discontinued from treatment with the study drug at any time due to unacceptable toxicity, disease progression and/or at the discretion of the investigator or the patient.

ELIGIBILITY:
Inclusion Criteria

Participants eligible for inclusion in this study must meet all of the following criteria:

1. Written informed consent must be obtained and signed prior to participation in the study
2. Male or female patients with a diagnosis of CML-CP ≥ 18 years of age
3. Patients must meet all of the following laboratory values at the screening visit:

   * < 15% blasts in peripheral blood and/or bone marrow
   * < 30% blasts plus promyelocytes in peripheral blood and/or bone marrow
   * < 20% basophils in the peripheral blood
   * ≥ 50 x 109/L (≥ 50,000/ mm3) platelets
   * Transient prior therapy related thrombocytopenia (< 50,000/mm3 for ≤ 30 days prior to screening) is acceptable
   * No evidence of extramedullary leukemic involvement, with the exception of hepatosplenomegaly
4. Mutation Analysis testing performed 6 months before study entry
5. Prior treatment with a minimum of:

   * 2 prior ATP-site TKIs (i.e. imatinib, nilotinib, bosutinib, dasatinib or ponatinib) in case of absence of T315I mutation
   * 1 prior ATP site TKI (i.e. imatinib, nilotinib, bosutinib, dasatinib or ponatinib) in case of presence of T315I mutation
6. Failure (adapted from the 2020 ELN Recommendations) or intolerance to the most recent TKI therapy at the time of screening

   * Failure for CML-CP patients (CP at the time of initiation of last therapy) is defined as meeting at least one of the following criteria.
   * Three months after the initiation of therapy: >10% BCR-ABL1 on International Scale (IS) if confirmed within 1-3 months
   * Six months after the initiation of therapy: BCR-ABL1 ratio > 10% IS
   * Twelve months after initiation of therapy: BCR-ABL1 ratio > 1% IS
   * At any time after the initiation of therapy, loss of CHR, MR2
   * At any time after the initiation of therapy, the development of new BCR-ABL1 mutations which potentially cause resistance to current treatment
   * At any time 12 months after the initiation of therapy, BCR-ABL1 ratio ≥ 1% IS or loss of MMR
   * At any time after the initiation of therapy, new clonal chromosome abnormalities in Ph+ cells: CCA/Ph+
   * Intolerance is defined as:
   * Non-hematologic intolerance: Patients with grade 3 or 4 toxicity while on therapy, or with persistent grade 2 toxicity, unresponsive to optimal management, including dose adjustments (unless dose reduction is not considered in the best interest of the patient if response is already suboptimal)
   * Hematologic intolerance: Patients with grade 3 or 4 toxicity (absolute neutrophil count [ANC] or platelets) while on therapy that is recurrent after dose reduction to the lowest doses recommended by manufacturer
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2
8. Evidence of typical BCR-ABL1 transcript [e14a2 and/or e13a2] at the time of screening which are amenable to standardized RQ-PCR quantification.
9. Adequate end organ function, within 12 days before the first dose of asciminib treatment. Patients with mild to moderate renal and hepatic impairment are eligible if:

   * Total bilirubin ≤ 3.0 x ULN without AST/ALT increase
   * Aspartate transaminase (AST) ≤ 5.0 x ULN
   * Alanine transaminase (ALT) ≤ 5.0 x ULN
   * Serum lipase ≤ 1.5 x ULN. For serum lipase > ULN - ≤ 1.5 x ULN, value should be considered not clinically significant and not associated with risk factors for acute pancreatitis
   * Alkaline phosphatase ≤ 2.5 x ULN
   * Creatinine clearance ≥ 30 mL/min as calculated using Cockcroft-Gault formula
10. Patients must avoid consumption of grapefruit, Seville oranges or products containing the juice of each during the entire study and preferably 7 days before the first dose of study medications, due to potential CYP3A4 interaction with the study medications. Orange juice is allowed.
11. Treatment with medications that meet one of the following criteria is allowed if used with caution at least one week prior to the start of treatment with study treatment:

    * Moderate or strong inducers of CYP3A
    * Moderate or strong inhibitors of CYP3A
12. Patients must have the following electrolyte values (as per central laboratory tests) within normal limits or corrected to be within normal limits with supplements prior to first dose of study medication:

    * Potassium (potassium increase of up to 6.0 mmol/L is acceptable at study entry if associated with creatinine clearance within normal limits)
    * Total calcium (corrected for serum albumin); (calcium increase of up to 12.5 mg/dl or 3.1 mmol/L is acceptable at study entry if associated with creatinine clearance within normal limits)
    * Magnesium, with the exception of magnesium increase > ULN - 3.0 mg/dL; > ULN - 1.23 mmol/L associated with creatinine clearance (calculated using Cockcroft-Gault formula) within normal limits.

Exclusion Criteria:

Patients eligible for this study must not meet any of the following criteria:

1. Known second chronic phase of CML after previous progression to AP/BC
2. Previous treatment with a hematopoietic stem-cell transplantation
3. Cardiac or cardiac repolarization abnormality, including any of the following:

   * History within 6 months prior to starting study treatment of myocardial infarction (MI), angina pectoris, coronary artery bypass graft (CABG)
   * Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g., bifascicular block, Mobitz type II and third degree AV block)
   * QTcF at screening ≥450 msec (male patients), ≥460 msec (female patients)
   * Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:
   * Risk factors for Torsades de Pointes (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia
   * Concomitant medication(s) with a "Known risk of Torsades de Pointes" per wwwcrediblemeds.org/ that cannot be discontinued or replaced 7 days prior to starting study drug by safe alternative medication.
   * Inability to determine the QTcF interval
4. Severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol (e.g. uncontrolled diabetes, active or uncontrolled infection, pulmonary hypertension)
5. History of acute pancreatitis within 1 year of study entry or past medical history of chronic pancreatitis
6. Known presence of significant congenital or acquired bleeding disorder unrelated to cancer
7. History of other active malignancy within 3 years prior to study entry with the exception of previous or concomitant basal cell skin cancer and previous carcinoma in situ treated curatively
8. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection, or gastric bypass surgery)
9. Previous treatment with or known/ suspected hypersensitivity to asciminib or any of its excipients.
10. Participation in a prior investigational study within 30 days prior to randomization or within 5 half-lives of the investigational product, whichever is longer
11. Pregnant or nursing (lactating) women
12. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception.

    Highly effective contraception methods include:
    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy (with or without hysterectomy) total hysterectomy or bilateral tubal ligation at least six weeks before taking study treatment). In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening). The vasectomized male partner should be the sole partner for that subject.
    * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS) or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
    * In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
    * Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or bilateral tubal ligation at least six weeks before taking study medication. In the case of oophorectomy alone, women are considered post-menopausal and not of child bearing potential only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
13. Sexually active males unwilling to use a condom during intercourse while taking study treatment and for 3 days after stopping study (only for patients treated with asciminib). A condom is required for all sexually active male participants on asciminib treatment to prevent them from fathering a child AND to prevent delivery of study treatment via seminal fluid to their partner. In addition, these male participants must not donate sperm for the time period specified above.
14. If a patient is presenting with symptoms suggestive of possible COVID-19 infection, we advise ruling it out by appropriate testing recommended by health authorities.

    * Nucleic acid amplification tests for viral RNA (polymerase chain reaction), in order to measure current infection with SARS-CoV-2
    * Antigen tests for rapid detection of SARS-CoV-2
    * Antibody (serology) tests to detect the presence of antibodies to SARS-CoV-2

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2024-06-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Alaska Oncology and Hematology, Anchorage, Alaska
  - Arizona Oncology Associates, Phoenix, Arizona
  - Cancer Treatment Centers of America, Phoenix, Arizona
  - Pacific Shores Medical Group, Long Beach, California
  - Lundquist Inst BioMed at Harbor, Torrance, California
  - Rocky Mountain Cancer Centers, Boulder, Colorado
  - Memorial Cancer Institute, Hollywood, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Florida Cancer Specialists-North, St. Petersburg, Florida
  - Florida Cancer Specialists East, Stuart, Florida
  - Florida Cancer Specialists Pan, Tallahassee, Florida
  - Indiana Blood and Marrow Institute, Beech Grove, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Uni of Massachusetts Medical Center, Worcester, Massachusetts
  - Michigan Med University of Michigan, Ann Arbor, Michigan
  - Siteman Cancer Center, St Louis, Missouri
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Uni of Cincinnati Medical Center, Cincinnati, Ohio
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Northwest Cancer Specialists, Portland, Oregon
  - Texas Oncology, Dallas, Texas
  - Texas Oncology P A, Fort Worth, Texas
  - Univ of TX MD Anderson Cancer Cntr, Houston, Texas
  - Texas Oncology Northeast Texas, Tyler, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on
  https://www.clinicalstudydatarequest.com/

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2681

RESULTS

PARTICIPANT FLOW:
Period: Treatment Phase
Arm/Group | Cohort A | Cohort B | Cohort C
Started | 26 | 27 | 3
Treated (Safety Set) | 25 | 27 | 3
Completed | 12 | 20 | 0
Not Completed | 14 | 7 | 3
Not completed — Physician Decision | 9 | 3 | 3
Not completed — Adverse Event | 3 | 1 | 0
Not completed — Subject decision | 1 | 2 | 0
Not completed — Progressive disease | 0 | 1 | 0
Not completed — Enrolled but not treated and discontinued | 1 | 0 | 0
Period: Safety Follow-up Phase
Arm/Group | Cohort A | Cohort B | Cohort C
Started | 23 | 24 | 3
Completed | 20 | 23 | 3
Not Completed | 3 | 1 | 0
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Subject decision | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Cohort C | Total
Number analyzed (Participants) | 26 | 27 | 3 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 19 | 3 | 39
  >=65 years | 9 | 8 | 0 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 0 | 30
  Male | 10 | 13 | 3 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 1 | 7
  White | 21 | 22 | 1 | 44
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events and Serious Adverse Events for Cohorts A and B up to 24 Weeks
Description: Adverse events (AEs) and serious adverse events (SAEs) are summarized by cohort. Clinically significant findings for vitals, laboratory values and electrocardiogram (ECG) are reported as adverse events and or serious adverse events as determined by the investigator.
Time Frame: Baseline to up to 24 Weeks
Population: Safety set for cohorts A and B
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 25 | 27
Participants
  Adverse Events (AEs) | 23 | 26
  Serious Adverse Events (SAEs) | 1 | 3
  Fatal SAEs | 0 | 1
  AEs leading to treatment discontinuation | 2 | 1
  AEs leading to dose adjustment/interruption | 7 | 9

2. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events for Cohorts A, B and C by Week 48
Description: Adverse events (AEs) and serious adverse events (SAEs) were summarized by cohort. Clinically significant findings for vitals, laboratory values and electrocardiogram (ECG) were reported as adverse events and or serious adverse events as determined by the investigator.
Time Frame: Baseline up to 48 weeks
Population: Safety set (SS): all participants all who received at least one dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 25 | 27 | 3
Participants
  Adverse Events (AEs) | 24 | 26 | 3
  Serious Adverse Events (SAEs) | 2 | 3 | 1
  Fatal SAEs | 0 | 1 | 0
  AEs leading to treatment discontinuation | 3 | 1 | 0
  AEs leading to dose adjustment/interruption | 7 | 10 | 2

3. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events for Cohorts A, B and C by Week 72
Description: as for outcome 2
Time Frame: Baseline up to 72 weeks
Population: Safety set (SS): all participants all who received at least one dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 25 | 27 | 3
Participants
  Adverse Events (AEs) | 24 | 26 | 3
  Serious Adverse Events (SAEs) | 4 | 4 | 1
  Fatal SAEs | 0 | 1 | 0
  AEs leading to treatment discontinuation | 3 | 1 | 0
  AEs leading to dose adjustment/interruption | 8 | 11 | 2

4. Secondary Outcome: Percentage of Patients Achieving Complete Hematologic Response (CHR) for Cohorts A, B and C
Description: A complete hematologic response (CHR) is defined as all of the following present for ≥ 4 weeks:
  * White blood cell count (WBC) <10 x 10^9/L
  * Platelet count <450 x 10^9/L
  * Basophils <5%,
  * No blasts and promyelocytes in peripheral blood
  * Myelocytes + metamyelocytes < 5% in peripheral blood
  * No evidence of extramedullary disease, including spleen and liver
  The estimated cumulative incidence rates were presented.
Time Frame: Baseline to 12, 24, 48, 72 weeks
Population: Full Analysis Set (FAS): All participants to whom study medication had been assigned
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 26 | 27 | 3
Percentage of participants
  12 weeks | 76.9 [56.4 to 91.0] | 92.6 [75.7 to 99.1] | 100 [29.2 to 100]
  24 weeks | 76.9 [56.4 to 91.0] | 92.6 [75.7 to 99.1] | 100 [29.2 to 100]
  48 weeks | 76.9 [56.4 to 91.0] | 92.6 [75.7 to 99.1] | 100 [29.2 to 100]
  72 weeks | 76.9 [56.4 to 91.0] | 92.6 [75.7 to 99.1] | 100 [29.2 to 100]

5. Secondary Outcome: Percentage of Patients Achieving Major Molecular Response (MMR) for Cohorts A, B and C
Description: The rate of major molecular response (MMR) by 12, 24, 48 and 72 weeks after the start of first study medication is defined as ≥ 3 log reduction of BCR-ABL (transcript from standardized baseline or ≤0.1% BCR-ABL/ABL % by international scale, measured by real-time quantitative polymerase chain reaction (RQ-PCR). BCR-ABL fusion gene is also called the Philadelphia chromosome.
  The estimated cumulative incidence rates were presented.
Time Frame: Baseline up to 12, 24, 48, 72 weeks
Population: Full Analysis Set (FAS): All participants to whom study medication had been assigned
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 26 | 27 | 3
Percentage of participants
  12 weeks | 38.5 [20.2 to 59.4] | 44.4 [25.5 to 64.7] | 0 [0.0 to 70.8]
  24 weeks | 42.3 [23.4 to 63.1] | 63.0 [42.4 to 80.6] | 0 [0.0 to 70.8]
  48 weeks | 46.2 [26.6 to 66.6] | 70.4 [49.8 to 86.3] | 0 [0.0 to 70.8]
  72 weeks | 50.0 [29.9 to 70.1] | 70.4 [49.8 to 86.3] | 0 [0.0 to 70.8]

6. Secondary Outcome: Percentage of Patients Achieving Molecular Response (MR2) for Cohorts A, B and C
Description: The rate of molecular response (MR2) by 12, 24, 48 and 72 weeks after the start of first study medication is defined as ≥ 2 log reduction of BCR-ABL (transcript from standardized baseline or ≤ 1% BCR-ABL/ABL % by international scale, measured by real-time quantitative polymerase chain reaction (RQ-PCR). BCR-ABL fusion gene is also called the Philadelphia chromosome.
  The estimated cumulative incidence rates were presented.
Time Frame: Baseline up to 12, 24, 48, 72 weeks
Population: Full Analysis Set (FAS): All participants to whom study medication had been assigned
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 26 | 27 | 3
Percentage of participants
  12 weeks | 53.8 [33.4 to 73.4] | 70.4 [49.8 to 86.3] | 0 [0.0 to 70.8]
  24 weeks | 57.7 [36.9 to 76.7] | 85.2 [66.3 to 95.8] | 0 [0.0 to 70.8]
  48 weeks | 61.5 [40.6 to 79.8] | 85.2 [66.3 to 95.8] | 0 [0.0 to 70.8]
  72 weeks | 61.5 [10.6 to 79.8] | 85.2 [66.3 to 95.8] | 0 [0.0 to 70.8]

7. Secondary Outcome: Percentage of Patients Achieving Molecular Response 4 (MR4) for Cohorts A, B and C
Description: The rate of molecular response (MR4) by 12, 24, 48 and 72 weeks after the start of first study medication is defined as ≥ 4 log reduction of BCR-ABL (transcript from standardized baseline or ≤ 0.01% BCR-ABL/ABL % by international scale, measured by real-time quantitative polymerase chain reaction (RQ-PCR). BCR-ABL fusion gene is also called the Philadelphia chromosome.
  The estimated cumulative incidence rates were presented.
Time Frame: Baseline up to 12, 24, 48, 72 weeks
Population: Full Analysis Set (FAS): All participants to whom study medication had been assigned
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 26 | 27 | 3
Percentage of participants
  12 weeks | 30.8 [14.3 to 51.8] | 18.5 [6.3 to 38.1] | 0 [0.0 to 70.8]
  24 weeks | 30.8 [14.3 to 51.8] | 29.6 [13.8 to 50.2] | 0 [0.0 to 70.8]
  48 weeks | 38.5 [20.2 to 59.4] | 44.4 [25.5 to 64.7] | 0 [0.0 to 70.8]
  72 weeks | 38.5 [20.2 to 59.4] | 48.1 [28.7 to 68.1] | 0 [0.0 to 70.8]

8. Secondary Outcome: Percentage of Patients Achieving Molecular Response 4.5 (MR4.5) for Cohorts A, B and C
Description: The rate of molecular response (MR4.5) by 12, 24, 48 and 72 weeks after the start of first study medication is defined as ≥ 4.5 log reduction of BCR-ABL (transcript from standardized baseline or ≤ 0.0032% BCR-ABL/ABL % by international scale, measured by real-time quantitative polymerase chain reaction (RQ-PCR). BCR-ABL fusion gene is also called the Philadelphia chromosome.
  The estimated cumulative incidence rates were presented.
Time Frame: Baseline up to 12, 24, 48, 72 weeks
Population: Full Analysis Set (FAS): All participants to whom study medication had been assigned
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 26 | 27 | 3
Percentage of participants
  12 weeks | 23.1 [9.0 to 43.7] | 11.1 [2.4 to 29.2] | 0 [0.0 to 70.8]
  24 weeks | 26.9 [11.6 to 47.8] | 18.5 [6.3 to 38.1] | 0 [0.0 to 70.8]
  48 weeks | 30.8 [14.3 to 51.8] | 25.9 [11.1 to 46.3] | 0 [0.0 to 70.8]
  72 weeks | 30.8 [14.3 to 51.8] | 29.6 [13.8 to 50.2] | 0 [0.0 to 70.8]

9. Secondary Outcome: Time to Achieve CHR, MR2, MMR, MR4, MR4.5 for Cohorts A, B and C
Description: Time to achieving a response level is defined as the time from the date of the first dose of study medication to the first documented achievement of each defined response level. Time to achieve a specific response level was analyzed using the Kaplan-Meier Product-Limit method. Patients who are known to be without achieving that response level were censored at the last adequate assessment.
Time Frame: Baseline up to 72 weeks
Population: Full Analysis Set (FAS): All participants to whom study medication had been assigned
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 26 | 27 | 3
weeks
  CHR | 11.1 [11.1 to 12.00] | 11.9 [11.1 to 12.1] | 11.1 [10.9 to NA] — NA = not estimable as there were not enough events
  MMR | 24.0 [4.1 to NA] — NA = not estimable as there were not enough events | 22.9 [11.1 to 28.3] | NA [NA to NA] — NA = not estimable as there were not enough events
  MR2 | 8.3 [4.0 to 47.0] | 4.3 [3.9 to 11.6] | NA [NA to NA] — NA = not estimable s there were not enough events
  MR4 | 36.1 [11.1 to NA] — NA = not estimable as there were not enough events | 58.6 [23.1 to NA] — NA = not estimable as there were not enough events | NA [NA to NA] — NA = not estimable as there were not enough events
  MR4.5 | NA [23.1 to NA] — NA = not estimable as there were not enough events | NA [48.1 to NA] — NA = not estimable as there were not enough events | NA [NA to NA] — NA = not estimable as there were not enough events

10. Secondary Outcome: Duration of CHR, MR2, MMR, MR4 and MR4.5 for Cohorts A, B and C
Description: Duration of Response (DOR) is the time from the date of the first documented molecular response level to the date of first documented loss of the response level or death due to any cause, whichever occurs first. DOR for each response level was analyzed using the Kaplan-Meier Product-Limit method. Participants continuing without that event were censored at the date of their last adequate response assessment.
Time Frame: Baseline up 72 weeks
Population: All participants in the Full Analysis Set (FAS) who achieved a particular response. FAS: All participants to whom study medication had been assigned
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 20 | 25 | 3
weeks
  CHR | NA [NA to NA] — NA = not estimable as there were not enough events | NA [NA to NA] — NA = not estimable as there were not enough events | NA [NA to NA] — NA = not estimable as there were not enough events
  MMR: number analyzed (Participants) | 13 | 19 | 0
  MMR | NA [NA to NA] — NA = not estimable as there were not enough events | NA [NA to NA] — NA = not estimable as there were not enough events |
  MR2: number analyzed (Participants) | 16 | 23 | 0
  MR2 | NA [NA to NA] — NA = not estimable as there were not enough events | NA [NA to NA] — NA = not estimable as there were not enough events |
  MR 4: number analyzed (Participants) | 10 | 15 | 0
  MR 4 | NA [NA to NA] — NA = not estimable as there were not enough events | NA [2.9 to NA] — NA = not estimable as there were not enough events |
  MR 4.5: number analyzed (Participants) | 9 | 8 | 0
  MR 4.5 | NA [NA to NA] — NA = not estimable as there were not enough events | NA [NA to NA] — NA = not estimable as there were not enough events |

11. Secondary Outcome: Progression Free Survival (PFS) for Cohorts A, B and C
Description: Progression Free Survival (PFS) is defined as time from the first dose of study medication to disease progression to accelerated phase/blast crisis (AP/BC) or death due to any cause, whichever occurs first. PFS was analyzed using the Kaplan-Meier Product-Limit method. Subjects who did not progress were censored at the last adequate assessment.
Time Frame: Baseline up to 72 weeks
Population: Full Analysis Set (FAS): All participants to whom study medication had been assigned
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 26 | 27 | 3
weeks | NA [NA to NA] — NA = not estimable as there were not enough events | NA [NA to NA] — NA = not estimable as there were not enough events | NA [NA to NA] — NA = not estimable as there were not enough events

12. Secondary Outcome: Overall Survival Overall Survival (OS) for Cohorts A, B and C
Description: Overall Survival (OS) is defined as the time from the first dose of study medication to death due to any cause during study. If a patient was not known to have died, then OS was censored at the latest date the patient was known to be alive. OS was analyzed using the Kaplan-Meier Product-Limit method
Time Frame: Baseline up to 72 weeks
Population: Full Analysis Set (FAS): All participants to whom study medication had been assigned
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 26 | 27 | 3
weeks | NA [NA to NA] — NA = not estimable as there were not enough events | NA [NA to NA] — NA = not estimable as there were not enough events | NA [NA to NA] — NA = not estimable as there were not enough events

ADVERSE EVENTS:
Time Frame: From Baseline to 30 days after last treatment (up to a maximum of approximately 85 weeks).
Arm/Group | Cohort A | Cohort B | Cohort C
All-Cause Mortality (participants affected / at risk) | 0/25 | 2/27 | 0/3
Serious Adverse Events (participants affected / at risk) | 4/25 | 4/27 | 1/3
Other Adverse Events (participants affected / at risk) | 24/25 | 26/27 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=25) | Cohort B (N=27) | Cohort C (N=3)
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Oesophageal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 0
Pelvic infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Brain stem infarction (Nervous system disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=25) | Cohort B (N=27) | Cohort C (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0
Palpitations (Cardiac disorders) | 1 | 5 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 6 | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 6 | 0
Dry mouth (Gastrointestinal disorders) | 3 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 8 | 2
Vomiting (Gastrointestinal disorders) | 3 | 5 | 1
Fatigue (General disorders) | 10 | 9 | 1
Non-cardiac chest pain (General disorders) | 3 | 1 | 0
Oedema peripheral (General disorders) | 2 | 3 | 1
Peripheral swelling (General disorders) | 0 | 2 | 0
Pyrexia (General disorders) | 3 | 2 | 0
COVID-19 (Infections and infestations) | 8 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 2 | 0
Sinusitis (Infections and infestations) | 4 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 0
Viral diarrhoea (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 2 | 1
Amylase increased (Investigations) | 3 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 2 | 0
Lipase increased (Investigations) | 4 | 3 | 0
Neutrophil count decreased (Investigations) | 2 | 1 | 0
Platelet count decreased (Investigations) | 2 | 2 | 0
Weight increased (Investigations) | 2 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 5 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 4 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 10 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Dizziness (Nervous system disorders) | 3 | 3 | 0
Headache (Nervous system disorders) | 9 | 7 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 3 | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 2 | 1
Hot flush (Vascular disorders) | 1 | 1 | 1
Hypertension (Vascular disorders) | 4 | 5 | 0
Hypotension (Vascular disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-03-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT04666259/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-16): https://cdn.clinicaltrials.gov/large-docs/59/NCT04666259/SAP_001.pdf